CLINICAL TRIAL: NCT06639425
Title: Efficacy of Lactobacillus Paracasei LC19 on Newly Diagnosed Type 2 Diabetes
Brief Title: Efficacy of Lactobacillus Paracasei LC19 on Type 2 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Guang Wang, Director of Endocrinology, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-DM-Lp
Record Dates: First submitted 2024-10-05; First posted 2024-10-15 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactobacillus paracasei LC19 supplementation (Experimental)
  Interventions: Dietary Supplement: Lactobacillus paracasei LC19 supplementation
- Placebo probiotic milk powder (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo probiotic milk powder

INTERVENTIONS:
Dietary Supplement: Lactobacillus paracasei LC19 supplementation — Orally administered Lactobacillus paracasei LC19 strain product, in addition to lifestyle intervention. This product is a probiotic milk powder, and the Lactobacillus paracasei LC19 strain is capable of producing high levels of tryptophan-conjugated cholic acid (Trp-CA)( 25g/packet, 2 packets/day).
  Arms: Lactobacillus paracasei LC19 supplementation
Dietary Supplement: Placebo probiotic milk powder — Orally administered placebo probiotic milk powder, in addition to lifestyle intervention. The placebo probiotic strain also belongs to Lactobacillus paracasei species, but does not produce Trp-CA. These products have the same color, odor, appearance, and packaging (25g/packet, 2 packets/day).
  Arms: Placebo probiotic milk powder

SUMMARY:
This is a randomized, double-blind, placebo-controlled clinical trial. The objective of this trial is to determine whether Lactobacillus paracasei LC19 supplementation has a positive effect on glucose lowering in patients with type 2 diabetes (T2D).

DETAILED DESCRIPTION:
In this trial, approximately 60 drug-naive patients with newly diagnosed Type 2 Diabetes (T2D) will be recruited. Laboratory evaluations will be conducted on the subjects to confirm their eligibility before randomization. After the screening, eligible subjects will be randomly assigned in a 1:1 ratio to either the Lactobacillus paracasei LC19 supplementation group or the placebo group during the randomization visit. They will then enter a 12-week double-blind treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years, both genders eligible
* Drug-naive patients with newly diagnosed type 2 diabetes
* Subjects with screening HbA1c ≥ 7.0% and ≤ 9.0%
* Subjects understand the nature, significance, potential benefits, inconvenience, and risks and procedure of the study, and voluntarily sign the informed consent form

Exclusion Criteria:

* Other types of diabetes except T2D: type 1 diabetes (including adult latent autoimmune diabetes), special type diabetes, or secondary diabetes (such as acromegaly or Cushing&#39;s syndrome, etc.)
* Subjects with acute diabetic complications such as diabetic ketoacidosis or diabetic hyperosmolar coma in the past 6 months
* Subjects with history of hypoglycemia in the past 6 months
* Subjects with history of New York Heart Association class (NYHA) grade of heart function ≥ III or serious cardiovascular diseases (myocardial infarction, or with the history of cardiac interventional therapy or stent implantation, valve disease or valve repair, unstable angina, transient ischemic attack or stroke) within 6 months before the screening period
* Subjects with history of chronic active hepatitis and/or severe liver dysfunction, renal dysfunction, and thyroid dysfunction
* Subjects with a medical history of malignant tumor
* Subjects with history of gastrointestinal diseases that affect food digestion and absorption (such as severe diarrhea, constipation, irritable bowel syndrome, inflammatory bowel disease, active gastrointestinal ulcers, acute cholecystitis, etc.) or with a history of intestinal resection or other gastrointestinal surgery (such as cholecystectomy) within one year before the screening period
* Subjects with history of surgery, or severe trauma in the past 6 months, or planning to undergo surgery during the study period
* Subjects suffering from severe infections, severe anemia, or neutropenia
* Subjects pregnant or in lactation, or those planning to become pregnant or impregnate during or within 3 months after the study period
* Subjects with history of receiving immunosuppressants, steroids, anti diarrheal drugs, antibiotics, lipid-lowering drugs, or other gastrointestinal motility medications within the past 3 months;
* Subjects using other medications that can affect blood glucose in the past 3 months
* Subjects with consumption of other probiotic or prebiotic products in the past 3 months before secreening
* Subjects with lactose intolerance, known or suspected allergy to probiotics used in experiments, history of drug allergies or allergic diseases
* Subjects with weight fluctuations ≥ 5kg in the past 3 months or planning to take medication to control weight during the study period
* Subjects with history of mental illness or epilepsy, or taking antidepressant medications
* Subjects with history of alcohol abuse (for men, alcohol consumption exceeding 40 grams per day and for women, exceeding 20 grams per day)
* Subjects have participated in any other clinical study in the past 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-12 (Actual); Primary Completion 2026-10-14 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c change | From enrollment to the end of treatment at 12 weeks
  Changes in HbA1c from baseline at12 weeks during follow-up

SECONDARY OUTCOMES:
fasting blood glucose change | From baseline at 4, 8, and 12 weeks during follow-up
  Changes in fasting blood glucose from baseline at 4, 8, and 12 weeks during follow-up
Glycated albumin change | From baseline at 4 and 12 weeks during follow-up
  Changes in glycated albumin from baseline at 4 and 12 weeks during follow-up
Glycemic achieving rate | From enrollment to the end of treatment at 12 weeks
  Glycemic achieving rate with HbA1c<6.5% at 12-week follow-up
Glucose tolerance | From baseline at 4 and 12 weeks during follow-up
  Changes in blood glucose levels (at 0, 30, 60, and 120 minutes during OGTT) from baseline at 4 and 12 weeks during follow-up
Insulin change | From baseline at 4 and 12 weeks during follow-up
  Changes in insulin levels (at 0, 30, 60, and 120 minutes during OGTT) from baseline at 4 and 12 weeks during follow-up
Plasma GLP-1 change | From baseline at 4 and 12 weeks during follow-up
  Changes in GLP-1 levels (at 0, 30, 60, and 120 minutes during OGTT) from baseline at 4 and 12 weeks during follow-up
BMI change | From baseline at 4, 8, and 12 weeks during follow-up
  Changes in BMI from baseline at 4, 8, and 12 weeks during follow-up
Alteration of fecal metabolites | From enrollment to the end of treatment at 12 weeks
  Fecal metabolites analysis from baseline to 12-week follow-up
Alteration of gut microbiome | From enrollment to the end of treatment at 12 weeks
  Fecal metagenomics sequencing from baseline to 12-week follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Guang Wang, MD, Principal Investigator — Beijing Chao Yang Hospital
Locations (1):
- Beijing Chao-yang Hospital, Capital Medical University, Beijing, Beijing Municipality, China